CLINICAL TRIAL: NCT00839787
Title: The Effect of Opiate Administration in Children With Acute Abdominal Pain and Peritoneal Signs on the Decision for Surgical Intervention
Brief Title: The Effect of Pain Medication in Children With Acute Abdominal Pain and Its Implication Over the Surgeon's Decision
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll more patients
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 200901230503p
Record Dates: First submitted 2009-02-06; First posted 2009-02-10 (Estimated); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Abdominal Pain
MeSH Terms: conditions — Abdominal Pain | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Morphine (Experimental): Morphine Sulfate: If weight is <50 Kg; Morphine 0.1mg/kg IV to a maximum of 10mg can be given; if weight ≥ 50 Kg a maximum of 10mg can be given.
  Interventions: Drug: Morphine Sulfate
- Placebo (Placebo Comparator): Normal saline
  Interventions: Drug: Morphine Sulfate

INTERVENTIONS:
Drug: Morphine Sulfate — Morphine Sulfate group: If weight is <50 Kg; Morphine 0.1mg/kg IV to a maximum of 10mg can be given; if weight ≥ 50 Kg a maximum of 10mg can be given
  Other Names: Astramorph,Avinza,DepoDur,Duramorph,Infumorph,Kadian

SUMMARY:
Surgeons are the individuals who will operate on a patient if it is determined to be necessary after they present with abdominal pain. For that reason, the investigators want to study if giving a medicine (morphine) to children presenting to the ED with abdominal pain will alleviate pain without changing the patient's physical exam and the subsequent surgeon's decision.

The investigators also will record any side effects of morphine, any associated surgical complications, and to identify the ultimate diagnosis.

DETAILED DESCRIPTION:
Unfortunately, the current standard of care obviates the use of pain medication in children with acute abdominal pain while waiting for the attending pediatric surgeon to perform their examination and determine if the patient requires operative intervention. This process can sometimes be protracted.

This practice occurs currently because of the concerns that analgesia may alter physical findings, interfere with the diagnosis, and delay definitive surgical intervention resulting in increased morbidity. This point of view has been challenged recently.

We designed this study taking into account the paramount importance of the pediatric surgeon's role in determining the need for operative intervention in the ultimate management of patient's presenting with acute abdominal pain and signs and symptoms of peritonitis.

Our primary objective is to demonstrate that the administration of intravenous morphine will alleviate pain in children presenting to the Emergency Department (ED) with abdominal pain and peritoneal signs, without changing the patient's physical exam and the subsequent surgeon's operative decision.

Secondary objectives include recording any adverse events of morphine and associated surgical complications, and identification of the ultimate diagnosis.

This is a prospective, randomized double-blind, placebo-controlled clinical that will be conducted in the ED at Children's Medical Center of Dallas. Children aged 1 to 18 years with acute abdominal pain of ≤ 3 days duration, a moderate to severe pain score, and the presence of peritoneal signs will be eligible. Patients will be randomized to receive either 0.1mg/kg of intravenous morphine (maximum 10 mg) or an equal volume of placebo (0.9% saline).

An ED physician will obtain clinical data, determine the pain score, write a presumptive diagnosis and place an order for the study medication. A surgical physician will also obtain clinical data and write his/her disposition. This evaluation will be repeated at 30-120 minutes after administration of the study medication by the ED and surgical physicians.

Each subject will be monitored for 2 weeks after enrollment for follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 to18 years of age who present with acute abdominal pain and signs of peritoneal irritation of less than 5 days duration.
* Pain scores from moderate to severe
* Need for intravenous access and require surgical consultation.

Exclusion Criteria:

* Pregnancy
* Chronic pain (defined as pain of more than two weeks' duration). 3. Constipation (Bowel movement less than 3imes/week, hard, small, or difficult to eliminate)
* Prior abdominal surgery or traumatic abdominal pain.
* History of gastritis, peptic ulcer disease, gastro esophageal reflux disease.
* Chronic illnesses associated with pain such as Ulcerative colitis, Crohn's disease, sickle cell disease or altered perception to pain (autism, spina bifida, altered mental status).
* Previous use of morphine sulfate or other narcotic/medication known to alter pain
* Perception or mental status six hours prior to presentation in the ED.
* Prior allergy or anaphylaxis to morphine.
* Acute respiratory distress, hypotension (less than 5thpercentile for age).
* Renal, pancreatic or biliary disease

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To demonstrate that IV morphine will alleviate pain in children presenting to the Emergency Department with abdominal pain and peritoneal signs, without changing the patient's physical exam and the subsequent surgeon's operative decision. | 2 Hours post-medication

SECONDARY OUTCOMES:
Secondary objectives include recording any adverse events of morphine and associated surgical complications, and identification of the ultimate diagnosis. | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mercedes M Uribe, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Children's Medical Center at Dallas, Dallas, Texas, United States